CLINICAL TRIAL: NCT02772406
Title: Linked Color Imaging (LCI) Versus White Light for the Detection of Colorectal Dysplasia in Ulcerative Colitis
Brief Title: Linked Color Imaging vs. White Light for Colorectal Dysplasia in Ulcerative Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 307-LCI-003
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; colonoscopy; Dysplasia; Diagnosis
MeSH Terms: conditions — Colitis, Ulcerative; Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): (With LCI endoscopy and 1 month later with white light endoscopy) The patients will be evaluated by Linked Color Imaging and 1 month later evaluated by White Light endoscopy
  Interventions: Device: Linked Color Imaging
- Control group (Active Comparator): (With white light endoscopy and 1 month later with LCI endoscopy) The patients will be evaluated by White Light endoscopy and 1 month later evaluated by Linked Color Imaging
  Interventions: Device: white light imaging

INTERVENTIONS:
Device: Linked Color Imaging
  Arms: Experimental group
Device: white light imaging
  Arms: Control group

SUMMARY:
The purpose of the study is to determine whether a new colonoscopic viewing technique called Linked color imaging(LCI) helps endoscopists detect more dysplasia lesions in ulcerative colitis patients than conventional colonoscopy using white light alone.

DETAILED DESCRIPTION:
Patients with longstanding IBD have increased risk of colorectal cancer (CRC) compared to the general population. The association between duration of the disease and development of CRC is the rationale for endoscopic surveillance. Colonoscopic surveillance of ulcerative colitis patients has been shown to reduce the risk of colorectal cancer and allow detection at an earlier stage, but even with meticulous examination, some precancerous lesions or cancers are missed. The newly developed LCI system (FUJIFILM Co.) creates clear and bright endoscopic images by using short-wavelength narrow-band laser light combined with white laser light on the basis of BLI technology. LCI makes red areas appear redder and white areas appear whiter. Thus, it is easier to recognize a slight difference in color of the mucosa. This is a study to determine if using Linked color imaging (LCI) of the colon, rather than the usual white light on the colon, will improve the detection of more dysplasia lesions in ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:patients with ulcerative colitis who meet surveillance criteria Exclusion Criteria:pregnant patients,unable or unwilling to give informed consent,patients with severe active colitis who would be unsafe to endoscope

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The number of Colorectal Dysplasia detected by LCI | 6 months

SECONDARY OUTCOMES:
The endoscopic scores with LCI | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, M.D.,Ph.D., Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Leifeld L, Rogler G, Stallmach A, Schmidt C, Zuber-Jerger I, Hartmann F, Plauth M, Drabik A, Hofstadter F, Dienes HP, Kruis W; Detect Dysplasia Study Group. White-Light or Narrow-Band Imaging Colonoscopy in Surveillance of Ulcerative Colitis: A Prospective Multicenter Study. Clin Gastroenterol Hepatol. 2015 Oct;13(10):1776-1781.e1. doi: 10.1016/j.cgh.2015.04.172. Epub 2015 May 5. PMID 25952309
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/25952309